CLINICAL TRIAL: NCT03448276
Title: Immediate Effect Of Whole-Body Vibration And Walk Over Muscle Strength, Balance And Functional Performance In Elderly People With Osteoporosis And Osteopenia: Clinical Randomized Controlled Trial
Brief Title: Immediate Effect Of Whole-Body Vibration And Walk in Osteoporosis/Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria das Graças Rodrigues de Araújo, Professor, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vibration, Walk And Osteop; CAAE N. 80679117.5.0000.5208 (Other: UFPE)
Record Dates: First submitted 2018-02-02; First posted 2018-02-28 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Muscle Strength; Postural Balance; Vibration; Walking
MeSH Terms: conditions — Osteoporosis | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Two groups: The experimental group (GI) that will hold the training in the vibrating platform and the control group (GC) that will perform the walk, settling 1 treatment session.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple: a researcher shall be exclusively responsible for the evaluations and reevaluations not having knowledge of what intervention group the patient will enter. The patient will be allocated among three groups. After the final evaluations, all data will be analyzed by another researcher directed solely to that purpose. Therefore, there will be a triple blinding (researcher, patient and statistician).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training in the vibrating platform (Experimental): 20-minute workout will be held, which will include: heating (5 minutes and stretching for the muscles quadriceps and sural triceps), 10 and 5 min of cooling.
  Interventions: Other: Training in the vibrating platform
- Walk (Active Comparator): Will be held 30 minutes of training, which will include the heating (5 minutes of stretching for the muscles quadriceps and sural triceps), 10 and 5 min of cooling.
  Interventions: Other: Walk

INTERVENTIONS:
Other: Training in the vibrating platform — 20-minute workout will be held, which will include: heating (5 minutes and stretching for the muscles quadriceps and sural triceps), 10 and 5 min of cooling.
  Arms: Training in the vibrating platform
Other: Walk — Will be held 30 minutes of training, which will include the heating (5 minutes of stretching for the muscles quadriceps and sural triceps), 10 and 5 min of cooling.
  Arms: Walk

SUMMARY:
Introduction: Osteoporosis and Osteopenia are common bone disorders, characterized by low bone mass, signs of bone deterioration and are responsible for typical bone fragility. Physical activity is certainly a valid prevention tool because it contributes to a healthy energy balance, increasing muscle mass and providing beneficial effects in bone metabolism. Stress induced by more vigorous activities such as weight lifting, increases the risk of injury, particularly in the elderly. Therefore, alternative strategies with lower risk of injury are indicated such as whole body vibration and walk.

Objective: Compare the effect whole body vibration and walking on muscular strength, balance and functional performance in the elderly with Osteoporosis and Osteopenia

Methods: It is a clinical trial study, controlled, parallel, randomized and blind, which will follow the guidelines established in the Consolidated Standards of Reporting Trials (CONSORT). Participants will be randomly distributed in 2 groups: the experimental group (GI) that will hold the training in the vibrating platform and the control group (GC) that will perform the walk, settling 1 treatment session. All participants will be subjected to the initial and final assessment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of osteoporosis or osteopenia examination of bone densitometry;
* Patients without severe neurological disease, vascular disorders, labyrinthitis and blindness;
* No use of gait auxiliaries;
* No history of fractures of the lower limbs in the last year;
* Do not be an alcoholic inactive (0 to 5 points) or less active (6 to 11 points) accordance with the usual physical activity questionnaire (QAFH).

Exclusion Criteria:

-Patients who submit to hypertensive peak, nausea and dizziness during the training program.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Muscular strength | 20 minutes
  Test of 1 repetition maximum (1RM)
Balance | 20 minutes
  Berg Balance scale (BBS). Minimum score 0 and maximum 56, the lower the score the greater the risk of falls.
Functional performance | 20 minutes
  Timed Up and Go test (TUG)
Balance | 20 minutes
  Stabilometry by Baropodometry

SECONDARY OUTCOMES:
Plantar pressure distribution | 20 minutes
  Baropodometry

CONTACTS AND LOCATIONS:
Locations (1):
- UFPE, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No